CLINICAL TRIAL: NCT05259878
Title: Examining the Relationship Between Adverse Childhood Events and Chronic Pain in the Canadian Forces
Brief Title: Adverse Childhood Events Chronic Pain
Status: Suspended | Type: Observational
Why Stopped: Awaiting Approvals
Sponsor: Canadian Forces Health Services Centre Ottawa (Other)
Responsible Party: Principal Investigator, Gaurav Gupta, Principal Investigator, Canadian Forces Health Services Centre Ottawa
Other Study IDs: 2020-045
Record Dates: First submitted 2022-02-12; First posted 2022-03-02 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: A Control group of students at CFB Borden will be recruited to complete questionnaires.
  Interventions: Other: Adverse Childhood Events
- Patients with chronic pain: Patients are active service members, ranging from the age of 18-60 years old, referred primarily from the National Capital Region, CFB Petawawa, CFB Kingston, and CFB Trenton for consultation and management
  Interventions: Other: Adverse Childhood Events

INTERVENTIONS:
Other: Adverse Childhood Events — • The Adverse Childhood Events (ACE) scale is a validated 10-item binary questionnaire ("yes" or "no") that retrospectively measures domains of physical, emotional, and sexual abuse in the first 18 years of life. Scores range from 0 to 10 with higher scores indicating more adverse experiences during patients' childhood.

SUMMARY:
There is data to suggest that early childhood physical, emotional and sexual trauma could contribute to the development of chronic pain later in life, but this has not been studied in the Canadian Forces. The investigator will examine the relationship between adverse childhood events (ACE) and patient reported pain and function conducted within the CAF

DETAILED DESCRIPTION:
There is data to suggest that early childhood physical, emotional and sexual trauma could contribute to the development of chronic pain later in life, but this has not been studied in the Canadian Forces. The investigators will examine the relationship between adverse childhood events (ACE) and patient reported pain and function conducted within the CAF. Investigators therefore hypothesize that ACE scores will be independently associated with variation in physical limitations, pain intensity when compared with a control group that has no chronic pain.

Procedure Investigators will collect data on pain conditions, potential risk factors, and function using standard patient reported outcome measures. This data includes information about the patient occupation, pain conditions and impact on life, exercise levels, mood, childhood experiences, views on their condition and requests for care support.

Risks and risk mitigation Participation in this study is voluntary and therefore patients and controls could choose not to fill out surveys. They will also be made aware that they can withdraw consent at any time without having any effect on access to future medical care.

Investigators do not foresee significant associated risks but our consent form will also provide information on support resources should distress ensue. Patients' confidentiality/anonymity will be protected through multiple strategies.

The Physical Medicine and Rehabilitation clinic within the Canadian Forces Health Services Centre Ottawa services about 500 patients with complex chronic pain issues per year. Patients are active service members, ranging from the age of 18-60 years old, referred primarily from the National Capital Region, CFB Petawawa, CFB Kingston, and CFB Trenton for consultation and management. A Control group of students at CFB Borden will be recruited to complete questionnaires.

As the standard intake, patients will generally complete the patient reported outcome measures listed below. At that time, they will be made aware of the study by a member of the research team not involved in their care. The information handout included in Appendix H will be provided and posted in the clinic. Control patients without chronic pain, will be recruited by word of mouth and through the information handout.

Patient data compiled includes demographics consisting of age, gender, trade, pain conditions and comorbidities. Each patient will undergo a standard in-clinic assessment, which includes standard, validated patient reported outcome measures including body pain diagram, numeric pain scale (PEG), pain disability index (PDI), adverse childhood events (ACE), mood (PHQ-9), perceived injustice (IEQ) and exercise (IPAQ).

All questionnaires can be administered in English or French. Please see Appendix A.

Investigators have included various standardized and adapted versions of other questionnaires which will allow control for known confounders. Control participants will not fill out the litigation status form.

Investigators will complete an analysis of this data to determine the relationship between adverse childhood events and patient reported pain and functional status. A priori power analysis indicates that a sample of 136 patients would provide 90% statistical power, with α set at 0.05, to detect a medium effect size (f2 = 0.15) for a regression with five predictors if ACEs would account for 5% of the variability in physical function, and our complete model would account for 15% of the overall variability. To account for 5% incomplete responses, investigators will enroll 143 patients and 75 controls.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic pain and student controls providing consent to complete administered questionnaires

Exclusion Criteria:

* patients not willing or unable to provide consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The Physical Medicine and Rehabilitation clinic within the Canadian Forces Health Services Centre Ottawa services about 500 patients with complex chronic pain issues per year. Patients are active service members, ranging from the age of 18-60 years old, referred primarily from the National Capital Region, CFB Petawawa, CFB Kingston, and CFB Trenton for consultation and management. A Control group of students at CFB Borden will be recruited to complete questionnaires
Sampling Method: Non-Probability Sample
Enrollment: 193 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
The Adverse Childhood Events (ACE) scale | baseline
  A validated 10-item binary questionnaire ("yes" or "no") that retrospectively measures domains of physical, emotional, and sexual abuse in the first 18 years of life. Scores range from 0 to 10 with higher scores indicating more adverse experiences during patients' childhood.

SECONDARY OUTCOMES:
Pain, Enjoyment and General Activity Scale (PEG) | baseline
  a 3-question scale with scores from 0-10 looking to describe the change (if any) in activity limitations, symptoms, emotions and overall quality of life, related to the pain condition. Higher scores indicate poorer pain and function
The Pain Disability Index (PDI) | baseline
  to investigate the magnitude of self-reported pain-related disability, independent from region of pain or pain-related diagnosis. The items of the questionnaire are assessed on a 0-10 numeric rating scale in which 0 means no disability and 10 is maximum disability.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Canadian Forces Health Services Centre, Ottawa, Ontario
  - Canadian Forces Health Services-, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No